CLINICAL TRIAL: NCT02478255
Title: Longitudinal MR Imaging of Pulmonary Function in Patients Receiving Thoracic Radiation Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bastiaan Driehuys (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Bastiaan Driehuys, Associate Professor of Radiology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00059856; 1R01HL105643-01 (NIH)
Record Dates: First submitted 2015-06-16; First posted 2015-06-23 (Estimated); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-01

CONDITIONS: Radiation Injury
Keywords: Radiation induced lung injury; Xenon gas; hyperpolarized
MeSH Terms: conditions — Radiation Injuries

ARMS (2):
- Patients scheduled to undergo Radiation Therapy (RT) (Active Comparator): Patients scheduled to undergo Radiation Therapy (RT) for lung cancer, or other malignancies such as breast cancer or lymphoma that involve significant irradiation of the thoracic cavity.
  Interventions: Drug: Hyperpolarized 129-Xenon gas; Device: MRI
- Healthy volunteers (Active Comparator)
  Interventions: Drug: Hyperpolarized 129-Xenon gas; Device: MRI

INTERVENTIONS:
Drug: Hyperpolarized 129-Xenon gas — Hyperpolarized xenon will be administered in multiple doses in volumes up to 25% of subject total lung capacity (TLC) followed by a breath hold of up to 15 seconds. Subsequent 129Xe doses will only be administered once the subject is ready to proceed.
  Other Names: Hyperpolarized 129Xe
Device: MRI — Conventional 1H MRI will be used to provide anatomical reference scans, as well as pulmonary perfusion.

SUMMARY:
The purpose of this study is to determine whether magnetic resonance imaging (MRI) using inhaled hyper polarized xenon-129 (129Xe) gas, and conventional contrast can help visualize impaired lung function and detect changes over time in patients receiving treatment as well as those who don't. 129Xe is a special type of xenon gas and when inhaled during MRI may be able to show areas of abnormal thickening of parts of the lungs. These images combined with images taken with injected contrast agents or other special types of MRI such as conventional proton (1H) MRI may provide a better way to look at lung structure and function. The ultimate goal is to predict the degree of radiation-induced lung injury that will develop in a given patient for a given treatment plan. The investigators anticipate that these images will provide more specific information about lung disease than standard lung function tests. The use of 129Xe MRI is investigational. Investigational means that these tests have not yet been approved by the US Food and Drug Administration and are only available in research studies like this one. In addition, standard MRI with contrast is not typically done as standard of care for monitoring changes due to thoracic radiation therapy, therefore, its use in this study is also considered investigational.

Healthy volunteers are being asked to participate in this study because to develop a database of functional images that are representative of healthy lungs.

ELIGIBILITY:
Inclusion Criteria for Patients:

1. Patient scheduled to undergo thoracic RT at Duke University to a dose of at least 20 Gy
2. Willing and able to give informed consent and adhere to visit/protocol schedules

Exclusion Criteria for Patients:

1. Subject is less than 18 years old
2. MRI is contraindicated based on responses to MRI Screening questionnaire
3. Subject is pregnant or lactating
4. Respiratory illness of a bacterial or viral etiology within 30 days of MRI
5. Subject has any form of known cardiac arrhythmia
6. Subject does not fit into 129Xe vest coil used for MRI
7. Subject cannot hold his/her breath for 15 seconds
8. Subject deemed unlikely to be able to comply with instructions during imaging
9. Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Inclusion/Exclusion Criteria for Healthy Volunteers

1. Subject meets all criteria above but does not have a clinical diagnosis of respiratory disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Mammarappallil, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Scheduled to Undergo Radiation Therapy (RT) | Healthy Volunteers
Started | 17 | 8
Completed | 9 | 8
Not Completed | 8 | 0
Not completed — Physician Decision | 6 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Scheduled to Undergo Radiation Therapy (RT) | Healthy Volunteers | Total
Number analyzed (Participants) | 17 | 8 | 25
Age, Continuous [Mean (Full Range); unit: years] | 64.4 [48 to 87] | 34 [19 to 70] | 54.7 [19 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 12 | 7 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 17 | 7 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 14 | 3 | 17
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulmonary Function, as Measured by Ventilation Defect Percentage (VDP)
Description: "Ventilation" is defined as the regional 129Xe airspace signal divided by the top 1% of 129Xe airspace signal (representing open-airway ventilation). A "Ventilation Defect" is defined as any region of lung where the Ventilation signal is more than 2 standard deviations below the mean Ventilation signal of healthy volunteer subjects' lungs. "Ventilation Defect Percentage", or VDP, is defined as the volume of a subject's Ventilation Defects divided by the volume of the subject's lung, multiplied by 100%.
Time Frame: Baseline, following radiation treatment (up to 3 months)
Population: Subjects that completed visit 1 and visit 2 (n=10) were analyzed. Not applicable to the healthy volunteers group.
Measure: Mean (Standard Error); unit: Ventilation Defect Percentage (VDP)
Arm/Group | Patients Scheduled to Undergo Radiation Therapy (RT) | Healthy Volunteers
Number analyzed (Participants) | 10 | 0
Ventilation Defect Percentage (VDP) | -2.20 (1.7) |
Statistical Analysis 1: Comparison: Patients Scheduled to Undergo Radiation Therapy (RT); Test type: Other; p = 0.22, t-test, 2 sided

2. Secondary Outcome: Change in Gas Exchange Defect Percentage (EDP) Following RT (Radiation Treatment)
Description: "Gas exchange" is defined as the ratio of the signal from 129Xe transiently bonding with hemoglobin in the pulmonary capillaries to the local 129Xe airspace signal. In other publications, the investigators have referred to this as "RBC (red blood cell) transfer". A "Gas Exchange Defect" is defined as any region of lung where the Gas Exchange signal is more than 2 standard deviations below the mean Gas Exchange signal of healthy volunteer subjects' lungs. "Gas Exchange Defect Percentage", or EDP, is defined as the volume of a subject's Gas Exchange Defects divided by the volume of the subject's lung, multiplied by 100%.
Time Frame: Baseline, following RT (up to 3 months)
Population: Subjects that competed visit 1 and visit 2 (n=10) were analyzed. Not applicable to the healthy volunteers group.
Measure: Mean (Standard Error); unit: Gas Exchange Defect Percentage (EDP)
Arm/Group | Patients Scheduled to Undergo Radiation Therapy (RT) | Healthy Volunteers
Number analyzed (Participants) | 10 | 0
Gas Exchange Defect Percentage (EDP) | 5.20 (2.6) |

3. Secondary Outcome: RBC (Red Blood Cell) to Barrier Ratio Following RT
Description: "RBC:barrier ratio" is defined as the ratio of the whole lung signal from 129Xe transiently bonding with hemoglobin in the pulmonary capillaries to the whole lung signal from 129Xe in the alveolar barrier tissue.
Time Frame: Baseline, following RT (up to 3 months)
Population: Subjects that competed visit 1 and visit 2 (n=10) were analyzed. Not applicable to the healthy volunteers group.
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Patients Scheduled to Undergo Radiation Therapy (RT) | Healthy Volunteers
Number analyzed (Participants) | 10 | 0
Ratio | -0.021 (0.016) |

4. Secondary Outcome: Change in High Barrier Uptake Percentage (HBUP) Following RT
Description: "Barrier Uptake" is defined as the ratio of the regional signal from 129Xe dissolved in the interstitial space within the alveolar walls to the regional signal from 129Xe in the adjacent airspaces. "High Barrier Uptake" is defined as any region of lung where the Barrier Uptake signal is more than 2 standard deviations above the mean Barrier Uptake signal of healthy volunteer subjects' lungs. "High Barrier Uptake Percentage", or HBUP, is defined as the volume of a subject's lung exhibiting High Barrier Uptake divided by the total volume of the subject's lung, multiplied by 100%.
Time Frame: Baseline, following RT (up to 3 months)
Population: Subjects that competed visit 1 and visit 2 (n=10) were analyzed. Not applicable to the healthy volunteers group.
Measure: Mean (Standard Error); unit: Interstitial space to alveolar walls (%)
Arm/Group | Patients Scheduled to Undergo Radiation Therapy (RT) | Healthy Volunteers
Number analyzed (Participants) | 10 | 0
Interstitial space to alveolar walls (%) | 5.0 (4.0) |

5. Other Pre Specified Outcome: Change in Perfusion Defect Percentage (PDP) Following RT
Time Frame: Baseline, following RT (up to 3 months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 24 hours after Xenon MRI
Arm/Group | Patients Scheduled to Undergo Radiation Therapy (RT) | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/8
Other Adverse Events (participants affected / at risk) | 0/17 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT02478255/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT02478255/ICF_001.pdf